CLINICAL TRIAL: NCT05996380
Title: A Phase 1 Trial to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of SHR-3167 Single Injection in Healthy Subjects and Patients With Type 2 Diabetes
Brief Title: A Phase 1 Trial to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of SHR-3167 Single Injection in Healthy Subjects and Patients With Type 2 Diabetes
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHR-3167-101
Record Dates: First submitted 2023-08-02; First posted 2023-08-18 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-08

CONDITIONS: T2DM

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR-3167 (Experimental)
  Interventions: Drug: SHR-3167
- SHR-3167 Placebo (Placebo Comparator)
  Interventions: Drug: SHR-3167 Placebo

INTERVENTIONS:
Drug: SHR-3167 — SHR-3167, Single administration
  Arms: SHR-3167
Drug: SHR-3167 Placebo — SHR-3167 Placebo Single administration
  Arms: SHR-3167 Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, single-dose escalation trial was designed. There are 6 dose groups and 1 optional dose group: 0.5 mg, 2 mg, 8 mg, 25mg, 50 mg, 100 mg and 150 mg (optional). Eight healthy adult subjects or T2DM patients in each dose group (except for 0.5 mg dose group, only 4 subjects will be enrolled) are randomly assigned to subcutaneously injection of SHR-3167 or placebo according to 3:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 years ≤ age ≤ 55 years (healthy subjects) or 18 years ≤ age ≤ 65 years (T2DM patients)
2. 18.5 kg/m2≤ Body mass index (BMI) <26.0 kg/m2 (healthy subjects) or 18.5 kg/m2≤ BMI <35.0kg/m2 (T2DM patients), and male weight ≥50kg and female weight ≥45kg
3. T2DM patients: 7.0% ≤ HbA1c ≤9.5%, 7.5mmol/L≤ fasting blood glucose ≤15mmol/L
4. Healthy subjects: 3.9 mmol/L< fasting blood glucose < 6.1mmol/L and HbA1c ≤6.0% at screening
5. Signed and dated informed consent indicating that the subject has been informed of all pertinent aspects of the study.

Exclusion Criteria:

1. History of significant multiple and/or severe drug allergies or with a known allergy to the trial product or any medicine chemically related to the trial product
2. Presence of cancer or any clinically significant cardiac, respiratory, metabolic, renal, hepatic, gastrointestinal, endocrinological, dermatological, venereal, hematological, neurological, or psychiatric diseases or disorders.
3. History of severe cardiovascular and cerebrovascular disease, including heart failure (NYHA class II to IV), myocardial infarction, unstable angina pectoris, stroke or transient ischemic attack, severe arrhythmia, or coronary artery bypass grafting or percutaneous coronary intervention, 6 months before screening to before randomization;
4. T2DM patients:

   a) Severe hypoglycemia, frequent hypoglycemia, ketoacidosis, or hypertonic coma from 6 months before screening to before randomization; b) Known proliferative diabetic retinopathy ordiabetic macular edema, or non-proliferative diabetic retinopathy requiring treatment during the trial;
5. Those who had a severe infection, severe trauma, or had undergone surgery in the 12 weeks prior to screening, or planned to undergo surgery during the trial
6. Participants who participated in a clinical trial of any other drug or medical device from 3 months prior to screening to before randomization or planned to participate during the study period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2023-06-09 (Actual); Primary Completion 2024-01-25 (Estimated); Study Completion 2024-04-28 (Estimated)

PRIMARY OUTCOMES:
Safety endpoints: Number of Adverse Events | Start of Treatment to end of study (approximately 92 days)
  A summary of adverse events, including Serious Adverse Events(SAEs)

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Province Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided